CLINICAL TRIAL: NCT04304534
Title: Multicenter, Randomized, Placebo Controlled, Double-blind, Parallel Group, Dose-finding Phase 2 Study to Evaluate the Efficacy and Safety of BAY 2433334 in Patients Following an Acute Myocardial Infarction
Brief Title: Study to Gather Information About the Proper Dosing and Safety of the Oral FXIa Inhibitor BAY 2433334 in Patients Following an Acute Heart Attack
Acronym: PACIFIC-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20603; 2019-003244-79 (EudraCT Number)
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY 2433334 high dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY 2433334 medium dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY 2433334 low dose (Experimental)
  Interventions: Drug: BAY2433334
- BAY2433334 matching placebo (Placebo Comparator)
  Interventions: Other: BAY2433334 matching placebo

INTERVENTIONS:
Drug: BAY2433334 — Tablet, taken orally once a day.
  Arms: BAY 2433334 high dose; BAY 2433334 low dose; BAY 2433334 medium dose
Other: BAY2433334 matching placebo — Tablet, taken orally once a day.
  Arms: BAY2433334 matching placebo

SUMMARY:
The purpose of this study is to try to find the best dose of the new drug BAY 2433334 to give to participants and to look at how well BAY 2433334 works on top of a dual antiplatelet therapy (acetylsalicylic acid +/- clopidogrel) in patients following a recent heart attack (myocardial infarction) that happens when a blood vessel in the heart suddenly becomes blocked. BAY 2433334, works by blocking a step of the blood clotting process in our body and thins the blood and is a so called oral FXIa inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 45 years of age or older, at the time of signing the informed consent
* Acute myocardial infarction (excluding MI associated with PCI or CABG revascularization procedures) with:

  * clinical symptoms of acute myocardial infarction AND
  * elevated biomarkers of myocardial necrosis (creatine kinase-muscle and brain isoenzyme [CK-MB] or cardiac troponins) AND
  * at least one of the following risk factors need to be fulfilled:

    * Age ≥ 65 years
    * Prior MI (before the index AMI event)
    * Prior peripheral arterial disease
    * Diabetes Mellitus
    * Prior coronary artery bypass grafting (CABG) AND
  * initial angiography and revascularization procedures, either PCI or CABG, as treatment for the index event performed before randomization. (Note: a planned, staged PCI procedure can be performed after randomization)
* Plan for dual antiplatelet therapy (ASA + P2Y12 inhibitor) after hospital discharge for the index AMI
* Randomization during hospitalization for the index AMI event and latest within 5 days of hospital admission
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent has to be signed before any study-specific procedure.

Exclusion Criteria:

* Hemodynamically significant ventricular arrhythmias or cardiogenic shock at time of randomization
* Active bleeding; known bleeding disorder, history of major bleeding (intracranial, retroperitoneal, intraocular) or clinically significant gastrointestinal bleeding within last 6 months of randomization
* Planned use or requirement of full dose and long term anticoagulation therapy during study conduct.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1601 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (160):
- United States (22):
  - Valley Clinical Trials, Inc. - Covina, Covina, California
  - Florida Premier Cardiology, Boynton Beach, Florida
  - Clearwater Cardiovascular Associates | Clearwater, FL, Clearwater, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - Southwest Florida Research, Naples, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Reid Health, Richmond, Indiana
  - Midwest Heart & Vascular Specialists, Overland Park, Kansas
  - Cardiovascular Associates Research, LLC, Covington, Louisiana
  - Southern Clinical Research, LLC, Zachary, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - White Oak Medical Center, Silver Spring, Maryland
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
  - Logan Health Research, Kalispell, Montana
  - Methodist Physicians Clinic, Omaha, Nebraska
  - The Valley Hospital, Inc., Ridgewood, New Jersey
  - Trinity Medical WNY, Cheektowaga, New York
  - Jefferson Heart Institute, Philadelphia, Pennsylvania
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - North Texas Research Associates, McKinney, Texas
- Austria (9):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt, Carinthia
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Medizinische Universität Graz, Graz, Styria
  - Krankenhaus St. Josef Braunau, Braunau am Inn, Upper Austria
  - Kepler Universitätsklinikum Campus III, Linz, Upper Austria
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Ottakring - Wilhelminenspital, Vienna
  - Klinik Floridsdorf - Krankenhaus Nord, Vienna
- Belgium (8):
  - OL Vrouwziekenhuis - Campus Aalst, Aalst
  - Imeldaziekenhuis - St-Elisabethkliniek, Bonheiden
  - AZ Sint-Jan Brugge-Oostende | Sint-Jan - Cardiology, Bruges
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - CHR de la Citadelle - Cardiology, Liège
- Czechia (11):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny, Brno
  - Nemocnice Ceske Budejovice, a.s. Department of kardiologie, České Budějovice
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
  - Fakultni nemocnice v Motole, Prague
  - Ustredni vojenska nemocnice Praha, Prague
  - Nemocnice Slany, Slaný
- Germany (10):
  - Universitätsherzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - St. Vinzenz-Hospital, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Sana-Klinikum Remscheid GmbH, Remscheid, North Rhine-Westphalia
  - Forschungszentrum Ruhr - KliFoCenter GmbH, Witten, North Rhine-Westphalia
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Krankenhaus Dresden-Friedrichstadt, Dresden, Saxony
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
- Hungary (11):
  - Allami Szivkorhaz, Balatonfüred
  - Budai Irgalmasrendi Korhaz, Budapest
  - University of Semmelweis/ Semmelweis Egyetem, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pandy Kalman Korhaz, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Josa Andras Hospital, Nyíregyháza
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz, Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (14):
  - A.O. San Pio, Benevento, Campania
  - ASL Caserta, Caserta, Campania
  - A.O.U. di Ferrara, Ferrara, Emilia-Romagna
  - Asl Roma 2, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Istituto Clinico Humanitas - Humanitas Mirasole S.p.A., Milan, Lombardy
  - IRCCS Centro Cardiologico Monzino S.p.A, Milan, Lombardy
  - ASST Valle Olona, Varese, Lombardy
  - A.O. S.Croce e Carle, Cuneo, Piedmont
  - ASL TO3 di Collegno e Pinerolo, Turin, Piedmont
  - A.O.U. di Sassari, Sassari, Sardinia
  - A.O.U. Ospedali Riuniti "Umberto I - G.M.Lancisi - G.Salesi", Ancona, The Marches
  - AUSL Toscana Sud-Est, Grosseto, Tuscany
  - ULSS3 Serenissima, Venezia, Veneto
- Japan (20):
  - Daido Hospital, Social Medical Corporation Kojunkai, Nagoya, Aichi-ken
  - Chiba-Nishi General Hospital, Matsudo, Chiba
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Hokkaido Cardiovascular Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji, Hyōgo
  - Takahashi Hospital, Kobe, Hyōgo
  - Nishinomiya Watanabe Cardiovascular Center, Nishinomiya, Hyōgo
  - Tsukuba Medical Center Hospital, Tsukuba, Ibaraki
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Shin-Kuki General Hospital, Kukichūō, Saitama
  - Saitama Sekishinkai Hospital, Sayama, Saitama
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku, Tokyo
  - Fukui Prefectural Hospital, Fukui
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Osaka General Medical Center, Osaka
  - Oita Prefectural Hospital, Ōita
- Netherlands (14):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noord West Ziekenhuisgroep-Medisch Centrum Alkmaar, Alkmaar
  - Reinier de Graaf Gasthuis, Delft
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Zuyderland Medisch Centrum, Heerlen
  - Elkerliek Ziekenhuis, Lokatie Helmond, Helmond
  - Leids Universitair Medisch Centrum, Leiden
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Ikazia Ziekenhuis, Rotterdam
  - VieCuri - Medisch Centrum voor Noord-Limburg locatie Venlo, Venlo
  - Gelre Ziekenhuizen Zutphen, Zutphen
  - Isala, Zwolle
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital sw. Wincentego a Paulo, Gdynia
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni, Grodzisk Mazowiecki
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Kliniczny Szpital Wojewodzki Nr 2 im. Sw. Jadwigi Krolowej, Rzeszów
  - Uniwersyteckie Centrum Kliniczne Warszawskiego UM, Warsaw
  - Szpital Grochowski im. dr.med. Rafala Masztaka, Warsaw
  - Uniwersytecki Szpital Kliniczny UM we Wroclawiu, Wroclaw
- Spain (12):
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i de Sant Pau | Cardiología, Barcelona
  - Hospital Universitari de Bellvitge | Bellvitge Biomedical Research Institute - Cardiology - AF, Stroke Prevention, Barcelona
  - Hospital Universitario Virgen de las Nieves|Cardiologia, Granada
  - Hospital Ramon y Cajal | Cardiologia, Madrid
  - Hospital Clinico Universitario San Carlos | Cardiologia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca | Neurology Department - Stroke, Murcia
  - Hospital Universitario Virgen de la Macarena, Seville
  - Inst Investigacio Sanitaria Pere Virgili | Hosp Univ Joan XXIII de Tarragona - Neurology - Stroke, No-Cardioembolic-Tia, Tarragona
  - Hospital Gral. Univ. de Valencia | Cardiologia, Valencia
  - Hospital Universitari i Politècnic La Fe | Cardiología, Valencia
- Sweden (9):
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Länssjukhuset Ryhov, Jönköping
  - Skånes Universitetssjukhus, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Danderyds sjukhus, Stockholm
  - Länssjukhuset Sundsvall-Härnösand, Sundsvall
  - Akademiska sjukhuset Hjärtforskningsmottagningen, Uppsala
  - Västmanlands Sjukhus Västerås, Västerås
- Switzerland (7):
  - Kantonsspital Baselland - Standort Liestal, Liestal, Basel-Landschaft
  - Kantonsspital Aarau, Aarau, Canton of Aargau
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Kantonsspital Baden, Baden
  - Hôpital Cantonal Universitaire de Genève, Geneva
  - Luzerner Kantonsspital, Lucerne
  - Ospedale regionale di Lugano, Lugano
- United Kingdom (5):
  - Lister Hospital, Stevenage, Hertfordshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Worcestershire Acute Hospital Trust, Worcester, Worcestershire
  - Imperial College London, London
  - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Whiteson HZ, Frishman WH. Factor XI/XIa Inhibitors: A New Approach to Anticoagulation. Cardiol Rev. 2025 Jul-Aug 01;33(4):306-311. doi: 10.1097/CRD.0000000000000624. Epub 2023 Dec 1. PMID 38038437
- [Derived] Rao SV, Kirsch B, Bhatt DL, Budaj A, Coppolecchia R, Eikelboom J, James SK, Jones WS, Merkely B, Keller L, Hermanides RS, Campo G, Ferreiro JL, Shibasaki T, Mundl H, Alexander JH; PACIFIC AMI Investigators. A Multicenter, Phase 2, Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Dose-Finding Trial of the Oral Factor XIa Inhibitor Asundexian to Prevent Adverse Cardiovascular Outcomes After Acute Myocardial Infarction. Circulation. 2022 Oct 18;146(16):1196-1206. doi: 10.1161/CIRCULATIONAHA.122.061612. Epub 2022 Aug 27. PMID 36030390
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 157 centers in 14 countries or regions, between 17-Jun-2020 (first participant first visit) and 21-Feb-2022 (last participant last visit)
Pre-assignment Details: 1664 participants were screened, 63 participants were screening failures. 1601 participants were randomized in a 1:1:1:1 ratio to 4 treatment groups: 397, 401, and 402 participants to the asundexian 10 mg, 20 mg and 50 mg groups and 401 participants to the placebo group
Groups:
- Asundexian 10 mg: Participants received Asundexian (BAY2433334) 10 mg
- Asundexian 20 mg: Participants received Asundexian (BAY2433334) 20 mg
- Asundexian 50 mg: Participants received Asundexian (BAY2433334) 50 mg
- Placebo: Participants received placebo
Period: Overall Study
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Started (Full analysis set (FAS)) | 397 | 401 | 402 | 401
Treated (Safety analysis set (SAF)) | 395 | 397 | 402 | 399
Completed | 303 (Treatment completed) | 317 (Treatment completed) | 309 (Treatment completed) | 309 (Treatment completed)
Not Completed | 94 | 84 | 93 | 92
Not completed — Subject decision COVID-19 pandemic related | 1 | 0 | 1 | 0
Not completed — Non-Compliance with study drug | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2 | 3
Not completed — Unspecific | 4 | 2 | 2 | 2
Not completed — Technical Problems | 2 | 2 | 3 | 4
Not completed — Death | 7 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 7 | 2 | 7 | 4
Not completed — Physician Decision | 4 | 9 | 9 | 5
Not completed — Subject Decision | 34 | 25 | 25 | 26
Not completed — Adverse Event | 35 | 40 | 39 | 44

BASELINE CHARACTERISTICS:
Population: FAS(Full data analysis)
Groups:
- Total: Total of all reporting groups
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo | Total
Number analyzed (Participants) | 397 | 401 | 402 | 401 | 1601
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 122 | 123 | 118 | 136 | 499
  >=65 years | 275 | 278 | 284 | 265 | 1102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 87 | 100 | 90 | 370
  Male | 304 | 314 | 302 | 311 | 1231
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 0 | 3
  Asian | 53 | 50 | 50 | 50 | 203
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 2 | 1 | 8
  White | 334 | 345 | 347 | 339 | 1365
  More than one race | 1 | 0 | 2 | 2 | 5
  Unknown or Not Reported | 5 | 2 | 1 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Number of Participants With Composite of CV Death, MI, Stroke and Stent Thrombosis (ST)
Description: CV death included death due to stroke, MI, heart failure or cardiogenic shock, sudden death or any other death due to other cardiovascular causes. Death due to non-traumatic hemorrhage was included.
  Acute MI was used when there was evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia.
  Stroke was defined as an acute episode of focal or global neurological dysfunction caused by an injury of the brain, spinal cord, or retina as a result of hemorrhage or infarction.
  ST was defined incorporating diagnostic certainty as well as timing: "Definite" ST: The highest level of certainty. Either angiographic or pathological confirmation of stent thrombosis. "Probable" ST: Regardless of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 27 | 24 | 22 | 22
Statistical Analysis 1: Comparison: Asundexian 20 mg vs Asundexian 50 mg vs Placebo; Comparison of the Asundexian 20 mg group and 50 mg group versus Placebo group; Test type: Other — HRs were only calculated if at least three events occurred in one of the compared groups and at least one event in each of the compared treatment groups. The competing event was non-CV death for events that include CV death; p = 0.8439, Log Rank; Cox Proportional Hazard = 1.052, 90% CI 2-sided [0.687 to 1.612]
Statistical Analysis 2: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.7562, Log Rank; Cox Proportional Hazard = 1.096, 90% CI 2-sided [0.674 to 1.781]
Statistical Analysis 3: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.978, Log Rank; Cox Proportional Hazard = 1.008, 90% CI 2-sided [0.614 to 1.656]

2. Primary Outcome: Safety - Number of Participants With BARC Bleeding Definition Type 2, 3 and 5
Description: Type 2: any overt, actionable sign of hemorrhage that doesn't fit the criteria for type 3 or 5 but meets at least one of the following criteria: 1) requires nonsurgical, med intervention by a HCP, 2) leads to hospital or rise in level of care, or 3) prompt eval. Type 3a: 1) overt bleed + Hg drop of 3 to <5 g/dl (provided Hg drop is related to bleed); 2 any transfusion with overt bleed. Type 3b: 1) overt bleed + Hg drop ≥5 g/dL (provided Hg drop is related to bleed); 2) cardiac tamponade; 3) bleed requiring surgical intervention for control (exclude dental/nasal /skin/hemorrhoid); 4) bleed requiring IV vasoactive agents. Type 3c: 1) ICH hemorrhage (doesn't include microbleeds or HT, does include intraspinal); subcategories confirmed by autopsy or imaging or LP; 2) intraocular bleed compromising vision. Type 5: fatal bleed. Type 5a: probable fatal bleed; no autopsy or image confirmation but clinical suspicion. Type 5b: definite fatal bleed; overt bleed or autopsy or image confirmation.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Asundexian: Asundexian 10 mg group and Asundexian 20 mg group and Asundexian 50 mg group
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo | Pooled Asundexian
Number analyzed (Participants) | 395 | 397 | 402 | 399 | 1194
Participants | 30 | 32 | 42 | 36 | 104
Statistical Analysis 1: Comparison: Placebo vs Pooled Asundexian; Comparison of the Pooled Asundexian group versus Placebo group; Test type: Other — HR was only calculated if at least three events occurred in one of the compared groups and at least one event in each of the compared treatment groups; p = 0.9158, Log Rank; Hazard Ratio (HR) = 0.98, 90% CI 2-sided [0.713 to 1.347]
Statistical Analysis 2: Comparison: Asundexian 10 mg vs Placebo; Comparison of the Asundexian 10 mg group versus Placebo group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.5633, Log Rank; Hazard Ratio (HR) = 0.867, 90% CI 2-sided [0.577 to 1.302]
Statistical Analysis 3: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.584, Log Rank; Hazard Ratio (HR) = 0.875, 90% CI 2-sided [0.587 to 1.306]
Statistical Analysis 4: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.417, Log Rank; Hazard Ratio (HR) = 1.202, 90% CI 2-sided [0.828 to 1.747]

3. Secondary Outcome: Efficacy - Number of Participants With CV Death
Description: CV death included death due to stroke, MI, heart failure or cardiogenic shock, sudden death or any other death due to other cardiovascular causes. Death due to non-traumatic hemorrhage was included.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 7 | 4 | 5 | 2
Statistical Analysis 1: Comparison: Asundexian 20 mg vs Asundexian 50 mg vs Placebo; Comparison of the Asundexian 20 mg group and Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.275, 90% CI 2-sided [0.322 to 5.050]
Statistical Analysis 2: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.991, 90% CI 2-sided [0.479 to 8.273]

4. Secondary Outcome: Efficacy - Number of Participants With MI
Description: Acute MI was used when there was evidence of myocardial necrosis in a clinical setting consistent with acute myocardial ischemia. According to MI Universal Definition from 2018 the diagnosis of MI requires combination of: 1. Presence of acute myocardial injury. 2. Evidence of acute myocardial ischemia derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery imaging, or in case of post-mortem pathological findings irrespective of biomarker values.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 18 | 20 | 18 | 17
Statistical Analysis 1: Comparison: Asundexian 20 mg vs Asundexian 50 mg vs Placebo; Comparison of the Asundexian 20 mg group and Asundexian 50 mg versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.125, 90% CI 2-sided [0.696 to 1.819]
Statistical Analysis 2: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other; Cox Proportional Hazard = 1.181, 90% CI 2-sided [0.686 to 2.031]
Statistical Analysis 3: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other — [test comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.070, 90% CI 2-sided [0.613 to 1.866]

5. Secondary Outcome: Efficacy - Number of Participants With Stroke
Description: Stroke was defined as an acute episode of focal or global neurological dysfunction caused by an injury of the brain, spinal cord, or retina as a result of hemorrhage or infarction.
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 4 | 3 | 0 | 2

6. Secondary Outcome: Efficacy - Number of Participants With Stent Thrombosis
Description: ST was defined incorporating diagnostic certainty as well as timing: "Definite" ST: The highest level of certainty. Either angiographic or pathological confirmation of stent thrombosis. "Probable" ST: Regardless of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 4 | 5 | 4 | 4

7. Secondary Outcome: Efficacy - Number of Participants With All Cause Mortality
Time Frame: From baseline up to 52 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 397 | 401 | 402 | 401
Participants | 10 | 7 | 10 | 7
Statistical Analysis 1: Comparison: Asundexian 20 mg vs Asundexian 50 mg vs Placebo; Comparison of the Asundexian 20 mg group and Asundexian 50 mg group versus Placebo group; Test type: Other — For all-cause mortality there is no competing event; p = 0.6016, Log Rank; Cox Proportional Hazard = 1.266, 90% CI 2-sided [0.603 to 2.658]
Statistical Analysis 2: Comparison: Asundexian 20 mg vs Placebo; Comparison of the Asundexian 20 mg group versus Placebo group; Test type: Other; p = 0.9945, Log Rank; Cox Proportional Hazard = 0.996, 90% CI 2-sided [0.414 to 2.401]
Statistical Analysis 3: Comparison: Asundexian 50 mg vs Placebo; Comparison of the Asundexian 50 mg group versus Placebo group; Test type: Other; p = 0.4085, Log Rank; Cox Proportional Hazard = 1.506, 90% CI 2-sided [0.667 to 3.405]

8. Secondary Outcome: Safety - Number of Participants With All Bleeding
Description: All bleeding events occurred from first intake of study intervention until 2 days after the last intake of study intervention
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 395 | 397 | 402 | 399
Participants | 70 | 75 | 82 | 85

9. Secondary Outcome: Safety - Number of Participants With BARC Bleeding Definition Type 3, 5
Description: Type 3a: 1) overt bleed + Hg drop of 3 to <5 g/dl (provided Hg drop is related to bleed); 2 any transfusion with overt bleed. Type 3b: 1) overt bleed + Hg drop ≥5 g/dL (provided Hg drop is related to bleed); 2) cardiac tamponade; 3) bleed requiring surgical intervention for control (exclude dental/nasal /skin/hemorrhoid); 4) bleed requiring IV vasoactive agents. Type 3c: 1) ICH hemorrhage (doesn't include microbleeds or HT, does include intraspinal); subcategories confirmed by autopsy or imaging or LP; 2) intraocular bleed compromising vision. Type 5: fatal bleed. Type 5a: probable fatal bleed; no autopsy or image confirmation but clinical suspicion. Type 5b: definite fatal bleed; overt bleed or autopsy or image confirmation.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 395 | 397 | 402 | 399
Participants | 5 | 3 | 3 | 5

10. Secondary Outcome: Safety - Number of Participants With BARC Bleeding Definition Type 1,2,3,5
Description: Type 1: bleeding that is not actionable and does not cause the patient to seek unscheduled performance of studies, hospitalization, or treatment by a healthcare professional; may include episodes leading to self-discontinuation of medical therapy by the patient without consulting a healthcare professional. For BARC bleeding definition 2,3 and 5, please refer to second primary endpoint.
Time Frame: From baseline up to 52 weeks
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
Number analyzed (Participants) | 395 | 397 | 402 | 399
Participants | 70 | 75 | 82 | 85

ADVERSE EVENTS:
Time Frame: After the first administration of study intervention for up to 52 weeks (but not starting after more than 2 days after the last administration). Reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, for up to 54 weeks.
Groups:
- Asundexian 10 mg: Subjects received Asundexian (BAY2433334) 10 mg for 26 weeks at least and up to 52 weeks
- Asundexian 20 mg: Subjects received Asundexian (BAY2433334) 20 mg for 26 weeks at least and up to 52 weeks
- Asundexian 50 mg: Subjects received Asundexian (BAY2433334) 50 mg for 26 weeks at least and up to 52 weeks
- Placebo: Subjects received Asundexian (BAY2433334) placebo for 26 weeks at least and up to 52 weeks
Arm/Group | Asundexian 10 mg | Asundexian 20 mg | Asundexian 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 10/397 | 7/401 | 10/402 | 7/401
Serious Adverse Events (participants affected / at risk) | 74/395 | 82/397 | 67/402 | 82/399
Other Adverse Events (participants affected / at risk) | 89/395 | 118/397 | 94/402 | 107/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 10 mg (N=395) | Asundexian 20 mg (N=397) | Asundexian 50 mg (N=402) | Placebo (N=399)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 9 (9) | 9 (12) | 10 (11) | 8 (8)
Angina pectoris (Cardiac disorders) | 5 (5) | 4 (4) | 6 (6) | 1 (1)
Angina unstable (Cardiac disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (5) | 4 (5) | 2 (2) | 5 (6)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interventricular septum rupture (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 5 (5) | 4 (4) | 4 (4)
Death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Vascular stent stenosis (General disorders) | 2 (2) | 2 (3) | 1 (1) | 2 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (2) | 7 (7) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coagulation factor VIII level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial bruit (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Von Willebrand's factor antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Von Willebrand's factor activity increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal epidural haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sigmoidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Revascularisation procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asundexian 10 mg (N=395) | Asundexian 20 mg (N=397) | Asundexian 50 mg (N=402) | Placebo (N=399)
Diarrhoea (Gastrointestinal disorders) | 22 (23) | 21 (22) | 22 (25) | 18 (19)
Chest pain (General disorders) | 13 (15) | 29 (32) | 15 (15) | 17 (20)
Dizziness (Nervous system disorders) | 18 (19) | 19 (22) | 21 (22) | 19 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 27 (28) | 21 (23) | 23 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (25) | 19 (45) | 21 (29) | 20 (26)
Hypertension (Vascular disorders) | 22 (23) | 27 (29) | 15 (15) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contracts Partners shall ensure that all patentable Results made by employees of Center or other parties involved by Contract Partners in connection with the performance of the Study, will be notified to Bayer without delay.

DOCUMENTS (2):
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04304534/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT04304534/SAP_001.pdf